CLINICAL TRIAL: NCT05980091
Title: Optimal Timing of Euploid Day 6 Blastocyst (blastocyst Which Was Biopsied on Day 6 After Fertilization) Transfer in Frozen Hormonal Replacement Therapy Cycles: Day 6 or Day 7 of Progesterone Administration?
Brief Title: Optimal Timing of Euploid Day 6 Blastocyst Transfer in Frozen HRT Cycles, Day 6 or Day 7 of Progesterone Administration.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ART Fertility Clinics LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2306-ABU-013-CC
Record Dates: First submitted 2023-07-25; First posted 2023-08-07 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-01

CONDITIONS: Infertility; Fertility Issues; Infertility, Female
Keywords: Implantation; Infertility; Blastocyst; HRT; Progesterone
MeSH Terms: conditions — Infertility; Infertility, Female | interventions — Estradiol; Progesterone; Embryo Transfer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Other): Embryo transfer is scheduled on the 6th full day of progesterone administration, following the initial commencement of progesterone (120 hours)
  Interventions: Diagnostic Test: Transvaginal ultrasound; Diagnostic Test: Serum LH, E2, P4; Drug: Estradiol Valerate 2 MG; Drug: Progesterone 100 Mg Vaginal Insert; Diagnostic Test: Serum P4 day of ET; Procedure: Embryo transfer
- Group B (Other): Embryo Transfer is scheduled on the 7th full day of progesterone administration, following the initial commencement of progesterone (144 hours)
  Interventions: Diagnostic Test: Transvaginal ultrasound; Diagnostic Test: Serum LH, E2, P4; Drug: Estradiol Valerate 2 MG; Drug: Progesterone 100 Mg Vaginal Insert; Diagnostic Test: Serum P4 day of ET; Procedure: Embryo transfer

INTERVENTIONS:
Diagnostic Test: Transvaginal ultrasound — Transvaginal ultrasound throughout the HRT cycle to not only monitor endometrial development but to also exclude the presence of an ovarian dominant follicle
Diagnostic Test: Serum LH, E2, P4 — In conjunction with ultrasound monitoring, participants will undergo serial measurements of serum Luteinizing Hormone (LH), Estradiol (E2) and Progesterone (P4) levels
Drug: Estradiol Valerate 2 MG — Participants will commence estradiol valerate 4 mg ( 2 x 2 mg) on day 2 / day 3 of menses.
  Estradiol will be increased to 6 mg on day 2 of estrogen treatment, and continued at a daily dose of 6 mg (3 tablets daily)
  Other Names: Estradiol Valerate
Drug: Progesterone 100 Mg Vaginal Insert — The initial progesterone dose of 100 mg will be commenced at 13hrs and repeated at 21hrs considered day 1 (vaginal suppository) when an optimal endometrial thickness for each participant has been achieved with a trilaminar appearance. The following day (day 2) progesterone administration will be increased to 100 mg vaginally three times daily
  Other Names: Progesterone 100 mg
Diagnostic Test: Serum P4 day of ET — On the day of embryo transfer (ET), a blood test is taken to measure serum P4
Procedure: Embryo transfer — Procedure in which embryo is transferred into the uterus
  Other Names: ET

SUMMARY:
The goal of this study is to compare the difference in clinical pregnancy, miscarriage and livebirth rate between day 6 euploid blastocyst transfer on the 6th and the 7th day of progesterone exposure in Hormonal Replacement Therapy (HRT) FET cycles. This prospective & randomized study will only include euploid day 6 blastocysts. This will be the first prospective study of euploid day 6 blastocysts thereby excluding aneuploidy as a cause of miscarriage and implantation failure. The point of randomization will occur on the day of progesterone commencement.

DETAILED DESCRIPTION:
Traditionally the duration of progesterone exposure before embryo transfer has been considered equal for day 5 and day 6 embryos but this may not be the case and warrants further study. The optimal preparation of the endometrium in frozen embryo transfer (FET) cycles is yet to be determined. Synchronization between the embryonic stage and the endometrial window of implantation (WOI) is crucial and progesterone plays a critical role in the WOI (1). Data on the optimal route of administration, the dose and duration of progesterone supplementation before blastocyst transfer are inconsistent (2,3). In view of the current lack of evidence, this study will be of importance.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years to 43 years.
* Having at least 1 euploid cryopreserved day 6 blastocyst of at least Grade BB quality.
* Endometrial trilaminar appearance on the day of progesterone start

Exclusion Criteria:

* Uterine abnormality
* Hydrosalpinx
* Asherman syndrome
* Any known contraindications or allergy to oral estradiol or progesterone.
* Intention to treat : exclusion factors :

  1. Spontaneous ovulation HRT cycle
  2. Discontinuation of HRT medication

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 316 (Estimated)
Dates: Start 2023-09-22 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Livebirth rate (LBR) | 41 weeks
  Defined as the delivery of a live infant born after 24 completed weeks of gestation

SECONDARY OUTCOMES:
Biochemical pregnancy rate | 5 weeks
  Positive hCG, but at 5 gestational weeks no ultrasonographic visible gestational sac seen but without a further development into a clinical pregnancy)
Clinical pregnancy rate | 5 weeks
  Ultrasonographic sac visible at 5 gestational weeks
Ongoing pregnancy rate after 12 weeks | 13 weeks
  Viable pregnancy with a gestational age of more than 12 weeks
Miscarriage rate | 24 weeks
  Spontaneous loss of a clinical pregnancy before 24 completed weeks of gestation

CONTACTS AND LOCATIONS:
Overall Officials: Carol Coughlan, PhD, Principal Investigator — ART Fertility Clinics LLC
Locations (2):
- United Arab Emirates (2):
  - ART Fertility Clinics LLC, Abu Dhabi, Abu Dhabi Emirate
  - ART Fertility Clinics Dubai, Dubai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Franasiak JM, Ruiz-Alonso M, Scott RT, Simon C. Both slowly developing embryos and a variable pace of luteal endometrial progression may conspire to prevent normal birth in spite of a capable embryo. Fertil Steril. 2016 Apr;105(4):861-6. doi: 10.1016/j.fertnstert.2016.02.030. PMID 26940791
- [Background] Nawroth F, Ludwig M. What is the 'ideal' duration of progesterone supplementation before the transfer of cryopreserved-thawed embryos in estrogen/progesterone replacement protocols? Hum Reprod. 2005 May;20(5):1127-34. doi: 10.1093/humrep/deh762. Epub 2005 Feb 3. PMID 15695314
- [Background] van de Vijver A, Drakopoulos P, Polyzos NP, Van Landuyt L, Mackens S, Santos-Ribeiro S, Vloeberghs V, Tournaye H, Blockeel C. Vitrified-warmed blastocyst transfer on the 5th or 7th day of progesterone supplementation in an artificial cycle: a randomised controlled trial. Gynecol Endocrinol. 2017 Oct;33(10):783-786. doi: 10.1080/09513590.2017.1318376. Epub 2017 Apr 26. PMID 28443690
- [Background] Zegers-Hochschild F, Adamson GD, Dyer S, Racowsky C, de Mouzon J, Sokol R, Rienzi L, Sunde A, Schmidt L, Cooke ID, Simpson JL, van der Poel S. The International Glossary on Infertility and Fertility Care, 2017. Fertil Steril. 2017 Sep;108(3):393-406. doi: 10.1016/j.fertnstert.2017.06.005. Epub 2017 Jul 29. PMID 28760517
- [Background] Roelens C, Santos-Ribeiro S, Becu L, Mackens S, Van Landuyt L, Racca A, De Vos M, van de Vijver A, Tournaye H, Blockeel C. Frozen-warmed blastocyst transfer after 6 or 7 days of progesterone administration: impact on live birth rate in hormone replacement therapy cycles. Fertil Steril. 2020 Jul;114(1):125-132. doi: 10.1016/j.fertnstert.2020.03.017. Epub 2020 Jun 16. PMID 32553469
- [Background] Bourdon M, Pocate-Cheriet K, Finet de Bantel A, Grzegorczyk-Martin V, Amar Hoffet A, Arbo E, Poulain M, Santulli P. Day 5 versus Day 6 blastocyst transfers: a systematic review and meta-analysis of clinical outcomes. Hum Reprod. 2019 Oct 2;34(10):1948-1964. doi: 10.1093/humrep/dez163. PMID 31644803
- [Background] Shapiro BS, Daneshmand ST, Garner FC, Aguirre M, Hudson C. Clinical rationale for cryopreservation of entire embryo cohorts in lieu of fresh transfer. Fertil Steril. 2014 Jul;102(1):3-9. doi: 10.1016/j.fertnstert.2014.04.018. Epub 2014 May 17. PMID 24842675